CLINICAL TRIAL: NCT05502588
Title: Effects of Forest Bathing and Environmental Factors on Individual Health Responses in Vancouver, B.C. Parks
Brief Title: Effects of Forest Bathing in Vancouver, B.C. Parks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, John Innes, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: H22-00216
Record Dates: First submitted 2022-08-03; First posted 2022-08-16 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Nature, Human; Mental Health Wellness 1; Stress, Psychological; Blood Pressure; Environmental Exposure; Anxiety
Keywords: Forest Bathing; Shinrin-yoku; Forest Therapy; Forest-based Intervention; Forest Immersion; Nature Therapy
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants are invited four times over one year to a forest bathing session that takes place on a barrier-free Vancouver, B.C. park trail. Each session is 2-hours including time for pre-test and post-test health measurements. At the study site participants will be randomized in 1:1 ratio to guided forest bathing walk or self-guided forest bathing walk. Subsequent sessions will be counterbalanced.
Who Masked: Participant
Masking Description: At the study site participants will be randomized in 1:1 ratio to guided forest bathing walk or self-guided forest bathing walk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Guided Forest Bathing (Active Comparator): Forest Bathing intervention without a guide and basic navigational instructions, explanation of forest bathing, and time to return.
  Interventions: Behavioral: Self-Guided Forest Bathing
- Guided Forest Bathing (Experimental): Forest Bathing intervention led by a certified Forest Therapy guide.
  Interventions: Behavioral: Guided Forest Bathing

INTERVENTIONS:
Behavioral: Self-Guided Forest Bathing — Participants will participate in two, 60-90 minute self-guided forest bathing sessions over the course of a year in one of four Vancouver, B.C. park trails and be given prompts to consciously use their five senses in the forest.
  Arms: Self-Guided Forest Bathing
Behavioral: Guided Forest Bathing — Participants will participate in two, 60-90 minute guided forest bathing sessions over the course of a year in one of four Vancouver, B.C. park trails. They will be invited by a certified forest therapy guide to consciously use their five senses in the forest.
  Arms: Guided Forest Bathing

SUMMARY:
This study aims to investigate environmental factors that influence people's responses to the Japanese practice of forest bathing in Vancouver, B.C. parks.

DETAILED DESCRIPTION:
The primary research aim is to investigate the relationship between biotic and abiotic factors in a sample of Vancouver, B.C. forested parks and specific health-related outcomes after forest bathing interventions. Forest bathing programs are a promising therapeutic method for enhancing heart rate and blood pressure functions and an effective psychological relaxation strategy. This study will investigate changes in autonomic nervous system activity and mood states after a 60-90 minute forest bathing program in four Vancouver, B.C. parks. Approximately 100 adult participants will be recruited for the study and participate in four sessions over one year. Physiological responses, pulse rate, systolic and diastolic blood pressure, and psychological indices will be measured before and after each session.

The health effects of forest-based interventions will vary due to environmental factors such as weather, temperature, humidity, light, and participants' psychological and physiological states. We are taking measurements pre- and post-treatment to detect any change in response during each session and seasonally.

Primary endpoint is to determine if the guided walk provides greater enhanced heart rate and blood pressure functions and an effective psychological relaxation strategy over the self-guided walk.

Secondary endpoints: 1) to determine if participants living in neighborhoods with below average street trees receive greater benefits than participants that live in neighborhoods with average or above average street trees, 2) assess changes within the same individuals over time 3) if there are different outcomes seasonally 4) if there are different outcomes between study sites.

ELIGIBILITY:
Inclusion Criteria:

* Adults (19+) that are residents of Vancouver, B.C.
* Spend time on a trail in a Vancouver park for at least 60 minutes per month
* Willing to refrain from tobacco products, alcohol, caffeine, marijuana, and psilocybin for at least two hours prior to arriving at the study site and during the forest bathing sessions

Exclusion Criteria:

* Must be able to move along a barrier-free trail independently
* Non-residents (e.g. tourists)
* Children (under 19 years of age)
* Participants with pets

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Abbreviated Profile of Mood States (POMS) - Change | Participants are tested before and after each forest bathing session and invited to attend four sessions during the study. Assessments for each session are included until the study ends. Forest bathing sessions will be held in 2022.
  Abbreviated Profile of Mood States (POMS) are routinely used by forest bathing researchers because psychologists regard it as rendering an accurate measure of mood states. The goal is to determine if spending time in a forest environment affects a psychological response. Abbreviated POMS contains 40 questions. Each answer is scored on a Likert Scale with values of 0, 1, 2, 3, and 4. Lower total scores indicated low mood problems, and conversely, a higher score may indicate a high mood problem. POMS will determine a baseline level of specific moods for a participant at the onset of the research trial and at the beginning and end of each forest bathing session.
Cardiovascular reactivity - Heart Rate - Change | Participants are tested before and after each forest bathing session and invited to attend four sessions during the study. Assessments for each session are included until the study ends. Forest bathing sessions will be held in 2022.
  Cardiovascular reactivity will be measured by participants taking heart rate before and after each forest bathing session.. Three measurements will be taken at 30-second intervals. The mean of the final two measurements taken for each interval will be used for statistical analysis.
Cardiovascular reactivity - Blood Pressure (Diastolic) - Change | Participants are tested before and after each forest bathing session and invited to attend four sessions during the study. Assessments for each session are included until the study ends. Forest bathing sessions will be held in 2022.
  Cardiovascular reactivity will be measured by participants taking diastolic blood pressure before and after each forest bathing session.. Three measurements will be taken at 30-second intervals. The mean of the final two measurements taken for each interval will be used for statistical analysis.
Cardiovascular reactivity - Blood Pressure (Systolic) - Change | Participants are tested before and after each forest bathing session and invited to attend four sessions during the study. Assessments for each session are included until the study ends. Forest bathing sessions will be held in 2022.
  Cardiovascular reactivity will be measured by participants taking systolic blood pressure before and after each forest bathing session. Three measurements will be taken at 30-second intervals. The mean of the final two measurements taken for each interval will be used for statistical analysis.

SECONDARY OUTCOMES:
Connectedness to Nature Scale (CNS) - Change | Participants are tested before and after each forest bathing session and invited to attend four sessions during the study. Assessments for each session are included until the study ends. Forest bathing sessions will be held in 2022.
  Connectedness to Nature Scale (CNS) is a scale designed to measure an individual's affective, experiential connection to nature. It was created based on the argument that for people to participate in environmental issues they need to feel part of the natural world. Another argument is that aspects of our urban or modern lifestyle relate to our nature connectedness and overall life satisfaction. The scale contains 13 items. It is a simple scale question with some reverse coded items Participants responded on a 5-point scale, where 1=strongly disagree and 5=strongly agree. CNS will determine a baseline level of nature relatedness and subjective well-being at the onset of the research trial and at the beginning and end of each forest bathing session.
Satisfaction With Life Scale (SWLS) - Change | Participants are tested before and after each forest bathing session and invited to attend four sessions during the study. Assessments for each session are included until the study ends. Forest bathing sessions will be held in 2022.
  The Satisfaction With Life Scale (SWLS) is a short 5-item instrument designed to measure global cognitive judgments of satisfaction with one's life.

CONTACTS AND LOCATIONS:
Overall Officials: John L. Innes, PhD, Principal Investigator — University of British Columbia
Locations (4):
- Canada (4):
  - Malcolm Knapp Research Forest, Maple Ridge, B.C.
  - Jericho Beach Park, Vancouver, B.C.
  - Pacific Spirit Regional Park, Vancouver, B.C.
  - Stanley Park, Vancouver, B.C.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UBC Forest Bathing Study Information and Consent Form — https://flex.redcap.ubc.ca/surveys/?s=9WXWAEEEWED7DWF7
- See also: John Innes, Professor, Faculty of Forestry — https://forestry.ubc.ca/faculty-profile/john-innes/